CLINICAL TRIAL: NCT03419481
Title: A Clinical Trial of Pembrolizumab in Patients with Hepatitis B Virus-related Hepatocellular Carcinoma, with Parallel Study on Baseline and Serial Change in the Immune Environment
Brief Title: Pembrolizumab in Hepatocellular Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CCTU (Other)
Responsible Party: Sponsor-Investigator, CCTU, Comprehensive Cancer Trial Unit, Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC053
Record Dates: First submitted 2018-01-10; First posted 2018-02-05 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: HCC
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- pembrolizumab (Experimental)
  Interventions: Drug: pembrolizumab

INTERVENTIONS:
Drug: pembrolizumab — 200mg every 3 weeks infusion

SUMMARY:
This is a single-arm Phase II trial of pembrolizumab in patients with hepatitis B virus-related hepatocellular carcinoma with parallel study on baseline and serial change in the immune environment.

Subjects should have a confirmed diagnosis of HCC (in accordance with the AASLD guideline) and confirmed chronic infection with hepatitis B virus as defined by positivity for HBsAg. Antiviral therapy for HBV must be given for at least 12 weeks and HBV viral load must be less than 100 IU/mL prior to first dose of study drug. They must have disease not amenable to a curative treatment approach or loco-ablation. Subject must be fit and agreeable with baseline and post-treatment biopsy of tumor. Subjects must have at least one measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, an Eastern Cooperative Oncology Group (ECOG) performance score of 0 or 1 and adequate organ functions. 30 subjects will be enrolled to receive pembrolizumab 200 mg IV every 3 weeks(Q3W). Pre-treatment and on-treatment biopsy after 2 cycles of Pembrolizumab will be preformed. Treatment will be stopped when progression of disease or intolerable toxicity occurs. The primary objectives of this trial are to study the efficacy and safety of pembrolizumab in patients with HBV-related HCC and to study the serial change in RNA expression of immune-related gene panel in post-treatment biopsy tissue.

The secondary objectives of this trial are to study the serial change in cytokine profile between pre-treatment and post-treatment samples, to study the PD-L1 immunohistochemical (IHC) expression in tumor sample at baseline and post-treatment tissue samples and to study the presence of tumor infiltrating lymphocytes in the baseline and post-treatment tumor samples.

The exploratory objective of this trial is to evaluate the possibility of using baseline and the serial change in RNA expression of immune-related gene panel or PD-L1/2 IHC to predict treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of advanced hepatocellular carcinoma (in accordance with the AASLD guidelines)
2. Confirmed chronic infection with hepatitis B virus as defined by positivity for HBsAg
3. For patients who are positive for HBsAg, antiviral therapy for HBV must be given for at least 12 weeks and HBV viral load must be less than 100 IU/mL prior to first dose of study drug. Subjects on active HBV therapy with viral loads under 100 IU/ml should stay on the same therapy throughout study treatment.
4. Disease extent is not amenable to curative surgery or loco-ablation
5. Patients who are fit and agreeable with baseline and post-treatment biopsy of tumor Subject Inclusion Criteria

   In order to be eligible for participation in this trial, the subject must:
6. Be willing and able to provide written informed consent/assent for the trial.
7. Be ≥ 18 years of age on day of signing informed consent.
8. Have measurable disease based on RECIST 1.1.
9. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor.
10. Have a performance status of 0 or 1 on the ECOG Performance Scale.
11. Demonstrate adequate organ function as defined, all screening labs should be performed within 10 days of treatment initiation.

    Adequate Organ Function Laboratory Values:

    Hematological Absolute neutrophil count (ANC) ≥1,200 /mcL Platelets ≥75,000 / mcL Hemoglobin ≥8g/dL without transfusion or EPO dependency (within 7 days of assessment) Renal Serum creatinine OR Measured or calculateda creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 X upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN Hepatic Serum total bilirubin ≤ 2mg/dL, or direct bilirubin≤ULN for those with total bilirubin > 2mg/dL or Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN AST (SGOT) and ALT (SGPT) ≤ 5 X ULN Albumin >3.0 mg/dL Coagulation International Normalized Ratio (INR) or Prothrombin Time (PT) orActivated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN Creatinine clearance should be calculated per institutional standard.
12. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
13. Female subjects of childbearing potential (Section 5.7.2) must be willing to use an adequate method of contraception as outlined in Section 5.7.2 - Contraception, for the course of the study through 120 days after the last dose of study medication.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
14. Male subjects of childbearing potential (Section 5.7.1) must agree to use an adequate method of contraception as outlined in Section 5.7.1- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapyor used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active TB (Bacillus Tuberculosis)
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Had a solid organ or hematologic transplant
6. Has had esophageal or gastric variceal bleeding within the last 6 months. All subjects will be screened for esophageal varices, unless such screening has been performed in the past 12 months before first dose of treatment. If varices are present, they should be treated according to institutional standards before starting trial treatment
7. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
8. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
9. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include cancer-insitu with curative treatment or malignancy more than 3 years prior to enrollment.
10. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
11. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
12. Has known history of, or any evidence of active, non-infectious pneumonitis.
13. Has an active infection requiring systemic therapy.
14. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
15. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
16. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
17. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
18. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
19. Has untreated active Hepatitis B Note: To qualify for enrollment, antiviral therapy for HBV must be given for at least 3 months, and HBV viral load must be less than 100 IU/mL prior to first dose of study drug. Those on active HBV therapy with viral loads under 100 IU/mL should stay on the same therapy throughout trial treatment. Those subjects who are anti-HBc (+), and negative for HBsAg, and negative for anti-HBs, and have an HBV viral load under 100 IU/mL do not require HBV anti-viral prophylaxis, but need close monitoring.
20. Baseline HBV DNA level > 100 IU/ml
21. Patients with concomitant HCV infection (as evidenced by Anti-HCV positivity)
22. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Response rate (RR) according to RECIST1.1 | 2 years

SECONDARY OUTCOMES:
1-year survival rate | 2 years
Response rate according to irRECIST | 2 years
Assessment of response duration | 2 years
Progression-free survival (PFS) | 2 years
Time-to-progression (TTP) | 2 years
Overall survival (OS) | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xiong Z, Chan SL, Zhou J, Vong JSL, Kwong TT, Zeng X, Wu H, Cao J, Tu Y, Feng Y, Yang W, Wong PP, Si-Tou WW, Liu X, Wang J, Tang W, Liang Z, Lu J, Li KM, Low JT, Chan MW, Leung HHW, Chan AWH, To KF, Yip KY, Lo YMD, Sung JJ, Cheng AS. Targeting PPAR-gamma counteracts tumour adaptation to immune-checkpoint blockade in hepatocellular carcinoma. Gut. 2023 Sep;72(9):1758-1773. doi: 10.1136/gutjnl-2022-328364. Epub 2023 Apr 5. PMID 37019619